CLINICAL TRIAL: NCT01410500
Title: Carfilzomib Multiple Myeloma Expanded Access Protocol for Patients With Relapsed and Refractory Disease
Status: Approved for marketing | Type: Expanded Access
Sponsor: Amgen (Industry)
Collaborators: Multiple Myeloma Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-002; NCT01495559 (obsolete NCT alias)
Record Dates: First submitted 2011-08-02; First posted 2011-08-05 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib was administered as an intravenous (IV) infusion over approximately 10 minutes on Days 1, 2, 8, 9, 15, and 16 of repeated 28-day cycles at a dose of 20 mg/m² on Days 1 and 2 of Cycle 1 and 27 mg/m² for all infusions thereafter until Cycle 12. For Cycle 13 and higher for those still receiving carfilzomib, the carfilzomib infusion schedule was abridged to Days 1, 2, 15, and 16 of each subsequent 28-day cycle. Carfilzomib treatment was continued until disease progression, diagnosis of a new malignancy, unacceptable toxicity, withdrawal of consent, or the study was terminated
  Other Names: Kyprolis®

SUMMARY:
The purpose of this study is to expand upon the safety data for carfilzomib by providing expanded access to patients with relapsed and refractory multiple myeloma who are unable to enroll in any other ongoing carfilzomib trial.

DETAILED DESCRIPTION:
This is a multi-center, expanded access, open label study of carfilzomib for patients with relapsed and refractory multiple myeloma. The study is designed to provide access to patients with relapsed and refractory disease that have received at least 4 prior regimens and are not eligible for any other enrolling carfilzomib Onyx-sponsored studies enrolling patients in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented multiple myeloma
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) status 0-2.
4. Life expectancy ≥ 3 months.
5. Measurable disease, defined as one or more of the following:

   * Serum M-protein ≥ 1 g/dL.
   * Urine M-protein ≥ 200 mg/24 hours.
   * For Immunoglobulin A (IgA) patients whose disease can only be reliably measured by serum quantitative immunoglobulin (qIgA), ≥ 750 mg/dl (0.75 g/dl).
6. For oligosecretory or non-secretory MM, either of the following:

   * Measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (ie, magnetic resonance imaging [MRI], computed tomography [CT] scan).
   * Documented abnormal free light chain ratio (NV: 0.26 to 1.65) or a value beyond the laboratory calculation range.
7. Received and either refractory or relapsed or discontinued due to toxicity to at least 4 prior lines of therapy as described below:

   * an immunomodulatory agent (lenolidamide or thalidomide)
   * bortezomib
   * an alkylating agent (standard or high dose)
   * a corticosteroid
8. Currently has progressive disease.
9. Refractory multiple myeloma defined as meeting one or more of the following:

   * Nonresponsive to most recent therapy (eg, stable disease only, or progressive disease while on treatment).
   * Disease progression within 60 days of discontinuation of most recent therapy (most recent therapy must be within 60 days of Screening).
10. Left ventricular ejection fraction (LVEF) ≥ 40% within 30 days before Cycle 1 Day 1. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation; multi gated acquisition scan (MUGA) is acceptable if ECHO is not available.
11. Adequate hepatic function, defined as aspartate aminotransferase (AST; SGOT) and alanine aminotransferase (ALT; SGPT) < 3 times the upper limit of normal and serum bilirubin ≤ 2.5 mg/dl.
12. Absolute neutrophil count ≥ 1,000 (may be supported by growth factors) and platelet count ≥ 40,000 within 14 days before Cycle 1 Day 1 without transfusion.
13. Creatinine clearance (CrCl) ≥15 mL/minute (measured or calculated using the Cockcroft and Gault Formula) within 14 days before Cycle 1 Day 1. This criterion does not apply to patients on hemodialysis.
14. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days before Cycle 1 Day 1 and must agree to use dual contraception methods for the duration of treatment and for 3 months following the last dose of treatment. Male patients must use an effective barrier method of contraception if sexually active with a female of childbearing potential during the treatment period and for 3 months following the last dose of treatment.
15. Written informed consent in accordance with federal, local, and institutional guidelines.

Exclusion Criteria:

1. Prior treatment with carfilzomib or enrollment in any other Phase 3 carfilzomib trial.
2. Known human immunodeficiency virus (HIV) seropositivity.
3. Active infection requiring systemic treatment with anti-biotics, anti-virals, or anti-fungals.
4. Known, active hepatitis A, B, or C viral infection.
5. Concomitant use of approved or investigational anti-cancer therapeutic agents, other than dexamethasone or palliative radiation therapy. Patients receiving radiation for pain control are eligible for enrollment in this study. No wash-out period is required for other anti-myeloma treatments received.
6. Concomitant use of other investigational agents (eg, anti-biotics or anti-emetics).
7. Pregnancy or breastfeeding.
8. History of plasma cell leukemia, defined as > 2.0 × 10ˆ9/L circulating plasma cells.
9. History of amyloidosis.
10. Known history of allergy to Captisol®.
11. Active congestive heart failure (New York Heart Association Class 3-4), symptomatic ischemia, conduction abnormalities uncontrolled by a conventional intervention, or a myocardial infarction within the past 4 months.
12. Intolerance to hydration due to pre-existing pulmonary, cardiac, or renal impairment. Patients on hemodialysis should be considered as meeting this criterion for entry.
13. Waldenström macroglobulemia or immunoglobulin M (IgM) myeloma.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen